CLINICAL TRIAL: NCT00313612
Title: A Phase II Study of Oxaliplatin Combined With Continuous Infusion Topotecan as Chemotherapy for Patients With Previously Treated Ovarian Cancer
Brief Title: Oxaliplatin and Topotecan in Advance Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00053; NYU 03-67 (Other: New York University); N01CM62204 (NIH)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2015-11-27 (Estimated); Last update posted 2015-11-27 (Estimated); Status verified 2013-05

CONDITIONS: Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Oxaliplatin; Topotecan; trioctyl phosphine oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (oxaliplatin plus topotecan) (Experimental): Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and topotecan IV continuously on days 1-14. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed at 30 days.
  Interventions: Drug: oxaliplatin; Drug: topotecan

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: topotecan — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO

SUMMARY:
This phase II trial is studying how well giving oxaliplatin together with topotecan works in treating patients with ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer. Drugs used in chemotherapy, such as oxaliplatin and topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the overall clinical response rate (complete and partial responses) in patients with previously treated ovarian epithelial, primary peritoneal, or fallopian tube cancer treated with oxaliplatin and topotecan.

II. Determine the toxic effects in patients treated with this regimen.

SECONDARY OBJECTIVES:

I. Estimate the time to progression and overall clinical response duration in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to response to prior platinum therapy (resistant vs sensitive).

Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and topotecan IV continuously on days 1-14. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ovarian epithelial, primary peritoneal, or fallopian tube cancer
* Meets 1 of the following criteria for response to prior platinum-based therapy:

  * Platinum-resistant disease, defined as a disease-free interval of < 6 months after prior platinum-based therapy OR progressive disease on a platinum-containing regimen
  * Platinum-sensitive disease, defined as a disease-free interval of > 6 months after prior platinum-based therapy
* Measurable or evaluable disease: Measurable disease is characterized as lesions reproducibly measurable in 1 dimension; evaluable disease is defined as known disease with CA125 levels > 50 U/mL on 2 occasions >= 1 week apart
* Previously treated with a taxane and platinum-based regimen, only 1 prior platinum-based regimen, including IV or intraperitoneal consolidation, one additional non-platinum and non-topotecan chemotherapy regimen allowed
* Life expectancy >= 4 months
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* AST =< 2.5 times ULN (5 times ULN if liver metastases are present)
* Creatinine =< 1.5 times ULN AND creatinine clearance > 40 mg/dL

Exclusion criteria:

* No presence of any other active cancer
* No uncontrolled intercurrent illness, including the following:

  * Infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No history of severe allergy to platinum compounds

  * (Mild reaction (skin only) allowed provided a negative skin test is obtained)
* No history of allergic reaction to appropriate antiemetics (e.g., 5HT3 antagonists)
* Recovered from prior chemotherapy
* At least 2 weeks since prior radiotherapy and recovered
* At least 4 weeks since prior investigational drugs
* No prior radiotherapy to the whole pelvic field
* No unresolved sequelae resulting from any surgical procedures
* No concurrent colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF]) during topotecan infusion
* No concurrent participation in another investigational trial
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-01; Primary Completion 2011-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - NYU Cancer Institute, New York, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Result] Stein SM, Tiersten A, Hochster HS, Blank SV, Pothuri B, Curtin J, Shapira I, Levinson B, Ivy P, Joseph B, Guddati AK, Muggia F. A phase 2 study of oxaliplatin combined with continuous infusion topotecan for patients with previously treated ovarian cancer. Int J Gynecol Cancer. 2013 Nov;23(9):1577-82. doi: 10.1097/IGC.0b013e3182a809e0. PMID 24172094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 39 patients were enrolled from 3 institutions between January 2006 and October 2009
Pre-assignment Details: 1 patient never received treatment
Groups:
- Treatment Stratum I (Oxaliplatin Plus Topotecan): Treatment stratum I (oxaliplatin plus topotecan) is resistant to prior platinum therapy. Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and topotecan IV continuously on days 1-14. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed at 30 days.
  oxaliplatin: Given IV
  topotecan: Given IV
- Treatment Stratum II (Oxaliplatin Plus Topotecan): Treatment stratum II (oxaliplatin plus topotecan) is sensitive to prior platinum therapy. Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and topotecan IV continuously on days 1-14. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed at 30 days.
  oxaliplatin: Given IV
  topotecan: Given IV
Period: Overall Study
Arm/Group | Treatment Stratum I (Oxaliplatin Plus Topotecan) | Treatment Stratum II (Oxaliplatin Plus Topotecan)
Started | 19 | 20
Completed | 19 | 19
Not Completed | 0 | 1
Not completed — Patient never received treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Stratum I: (Oxaliplatin Plus Topotecan): Treatment stratum I (oxaliplatin plus topotecan) is resistant to prior platinum therapy. Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and topotecan IV continuously on days 1-14. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed at 30 days.
  oxaliplatin: Given IV
  topotecan: Given IV
- Total: Total of all reporting groups
Arm/Group | Treatment Stratum I: (Oxaliplatin Plus Topotecan) | Treatment Stratum II (Oxaliplatin Plus Topotecan) | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Median (Full Range); unit: years] | 61 [38 to 80] | 59 [40 to 71] | 60 [38 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate (Complete and Partial Response by RECIST and/or CA [Cancer Antigen] 125)
Description: Tumor response was assessed every two cycles by CT/MRI using RECIST (Response Evaluation Criteria in Solid Tumors) criteria. Per Response Evaluation Criteria in Solid Tumors (RECIST 1.0) for target lesions: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >= 30% decrease in the sum of the longest diameter (LD) of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every two cycles for up to 24 weeks.
Population: 30 patients were analyzed. Eight patients discontinued treatment before 2 cycles.
Measure: Number; unit: participants
Groups:
- Treatment Stratum I (Oxaliplatin Plus Topotecan); Treatment Stratum II (Oxaliplatin Plus Topotecan): Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and topotecan IV continuously on days 1-14. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed at 30 days.
  oxaliplatin: Given IV
  topotecan: Given IV
Arm/Group | Treatment Stratum I (Oxaliplatin Plus Topotecan) | Treatment Stratum II (Oxaliplatin Plus Topotecan)
Number analyzed (Participants) | 16 | 14
participants
  Complete Response | 3 | 3
  Partial Response | 1 | 6
  Stable Disease | 8 | 4
  Disease Progression | 4 | 1

2. Secondary Outcome: Time to Disease Progression by RECIST and/or CA 125
Description: Time to disease progression by RECIST and/or CA 125
Time Frame: Tumor measurements will be performed every 8 weeks until the date of first documented progression up to 100 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Stratum I (Oxaliplatin Plus Topotecan) | Treatment Stratum II (Oxaliplatin Plus Topotecan)
Number analyzed (Participants) | 19 | 19
months | 6.3 [2.6 to 7.1] | 12.6 [4.3 to 16.2]

ADVERSE EVENTS:
Arm/Group | Treatment Stratum I (Oxaliplatin Plus Topotecan) | Treatment Stratum II (Oxaliplatin Plus Topotecan)
Serious Adverse Events (participants affected / at risk) | 14/19 | 12/19
Other Adverse Events (participants affected / at risk) | 18/19 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Stratum I (Oxaliplatin Plus Topotecan) (N=19) | Treatment Stratum II (Oxaliplatin Plus Topotecan) (N=19)
Neutropenia (Investigations) | 3 (3) | 12 (12)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
RBC transfusion (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombocytopenia (Investigations) | 5 (5) | 10 (10)
Platelet transfusion (Investigations) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Alanine aminotransferase (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Stratum I (Oxaliplatin Plus Topotecan) (N=19) | Treatment Stratum II (Oxaliplatin Plus Topotecan) (N=19)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (9) | 16 (16)
Anorexia (Metabolism and nutrition disorders) | 10 (10) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Weight loss (Investigations) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (9) | 18 (18)
Headache (Nervous system disorders) | 0 (0) | 5 (5)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less